CLINICAL TRIAL: NCT00870207
Title: Tu Salud Si Cuenta Worksite: Pilot Intervention Study
Acronym: TSSC Worksite
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Belinda Reininger, DrPH. - School of Public Health, University of Texas Health Science Center at Houston, Brownsville Regional Campus
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: HSC-SPH-09-0023; HSC-SPH-09-0023
Record Dates: First submitted 2009-03-26; First posted 2009-03-27 (Estimated); Last update posted 2011-05-03 (Estimated); Status verified 2011-04

CONDITIONS: Obesity; Physical Activity; Diet; Stress
Keywords: Feasibility of implementing TSSC in worksite environment
MeSH Terms: conditions — Obesity; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Immediate Intervention Group (Other): The immediate intervention group will receive the TSSC pilot worksite intervention in the initial 12 week period from the pre-test/enrollment visit.
  Interventions: Behavioral: Tu Salud Si Cuenta Worksite Intervention
- Delayed Intervention Group (Other): The delayed intervention group will receive the TSSC pilot worksite intervention beginning in month 6 of the study (6 months from the enrollment/pre-test visit).
  Interventions: Behavioral: Tu Salud Si Cuenta Worksite Intervention

INTERVENTIONS:
Behavioral: Tu Salud Si Cuenta Worksite Intervention — The intervention will consist of providing TSSC newsletters to employees of the worksite. Additionally, informational sessions about physical activity and healthful food choice (consistent with the TSSC messages) during work hours will be implemented. Social support groups for the behavior changes will be established thru colleague networks. Individualized behavior change plans will be designed for enrolled participants. Additionally, environmental changes including a well equipped exercise facility on site and access to healthful foods in vending machines and work groups providing fruit and vegetable access in kitchen area will be implemented.

SUMMARY:
Building on existing intervention strategies of the Tu Salud Si Cuenta media campaign, this proposed worksite pilot study will be testing a new feature by designing worksite promotion intervention strategies. The purpose of this study is to test the feasibility of a worksite-based physical activity and healthful food choice. The intervention will be among two worksites in the Lower Rio Grande Valley who employ primarily Mexican-American personnel.

DETAILED DESCRIPTION:
Obesity has not only been increasing over the past three decades (Wang & Beydoun, 2007; Wang & Zhang, 2002), it is predicted to increase in the future until by 2048 all American adults would be overweight (Wang, Beydoun, Liang, Caballero, Kumanyika, 2008). Moreover, the majority of Mexican American men and women are predicted to be overweight and obese by 2030 (91.1% and 86.7% respectively).

The proposed intervention research study is building from existing intervention strategies designed for the Mexican American population entitled Tu Salud Si Cuenta. This intervention highlights in the media successful role models who have changed their food choices and physical activity levels. In addition the intervention designs environmental changes to help community members carry out recommended behavior change strategies. Outcomes of interest for this study include increased physical activity so as to achieve the CDC/ACSM recommendations of 150 minutes of moderate to vigorous physical activity each week (Haskell et al., 2007), eating 5 servings of fruits and vegetables each day, reducing food portion sizes, and subsequent changes in biomarkers of health.

This proposed worksite pilot study will be testing a new feature to the TSSC intervention by designing worksite promotion intervention strategies to promote physical activity and healthful food choices through environmental change strategies at the worksite. The same full scope of behavioral and clinical outcomes of interest will be examined in this pilot.

The participants in this study will be male and female employees of two worksites, aged 18-65 years. A convenience sample will be used for this study. Employees from State Department of Public Health Region 11 Harlingen Office or City of Brownsville will be recruited. Supervisors from both sites have provided letters of support for this project and have agreed to allow recruitment. Employees will be contacted with informational flyers and e-mails sent by the supervisors providing the letters of support. Interested adults will be sent an interest letter and informed consent. Data collection will proceed after the participant completes the informed consent form and provides documentation of physician's clearance to participate in physical activity.

The purpose of this study is to test the efficacy of a worksite-based physical activity and healthful food choice, intervention among two worksites in the Lower Rio Grande Valley who employ primarily Mexican American personnel.

Persons will complete consent forms during an enrollment/pretest period of 4 weeks. This period will include an electronic pre-test survey using Survey Monkey online software (Finley, 2008) completed by each participant. Additionally, clinical measures such as blood pressure, anthropometrics, fasting total cholesterol, triglycerides and glucose will be collected for each participant. These exams will be conducted by the trained staff from the clinical research unit and follow the identical procedures used for members of the Hispanic Health Research Cohort. Finally, in line with the Centers for Disease Control and Prevention, each participant will be encouraged to visit their personal physician and discuss participation in the recommended 150 minutes of physical activity per week.

All individuals are given an exit interview with a registered phlebotomist or registered nurse to review immediate findings. All samples for laboratory testing and storage will be coded and identifiers removed. Participants will also provided with a written summary including their height, weight, waist circumference, blood pressure, fasting glucose, cholesterol and triglycerides. Values out of their expected range are flagged and referrals made as necessary. This interview is also used to address any questions or concerns that may be raised.

Descriptive analyses will be used to compare the characteristics of the participants in the intervention and control groups that we intend to compare with respect to any outcome of interests, (e.g., blood pressure). Specifically, we will compare the groups with respect to demographic and socio-economic factors such as age, sex, ethnicity, and education level. Since the outcome measurements at baseline and the follow up quarterly visit (at 3 months, 6 months, etc) are expected to be correlated, we will use Generalized Estimating Equations (GEE) models. GEE takes into account the correlation of an outcome measured repeatedly over time by treating it as a nuisance parameter (Zeger & Liang, 1986). As a result, the within-subjects correlation is not modeled explicitly. GEE uses a "working correlation" to treat the within-subjects correlation, and produces standard error estimates that take into account the correlation of responses with subjects. In addition, we will use Random effects models (Wolfinger & O'Connell, 1993) to adjust for the heterogeneity of subjects, which can be due to unmeasured predispositions, such as genetic factors, that account for the correlation within subjects across time. Estimated effects of a covariate of interest (e.g., males vs. females) are adjusted for these individual differences and model estimates should be interpreted in terms of the change due to the covariate in an individual at a given level of random subject effect. The random effects model is most useful when inferences about individual differences are the primary interest. Random effects models have been developed for both continuous and binary outcome variables (Wolfinger et al., 1993).

The study will take place over a 1 year time frame. Participants will have data collected prior to the intervention and four posttests at 3-month intervals. The immediate intervention group will receive the pilot worksite intervention for the initial 12 week period. The delayed intervention group will receive the pilot worksite intervention beginning in month 3 of the study.

ELIGIBILITY:
Inclusion Criteria:

* Men and women who are full- or part-time employees of either State Department of Public health Region 11 Harlingen Office or City of Brownsville.
* Persons of any racial/ethnic group aged between 18-65 years.
* Persons who are comfortable communicating in English (speaking, reading, and writing).
* Persons who are cleared by a physician for participation in the study.

Exclusion Criteria:

* Persons older than 65 years or younger than 18 years.
* Persons not currently employed with either of the two worksite partners.
* Persons who are not medically cleared by personal physician.
* Persons who are not comfortable communicating in English (speaking, reading, and writing).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2010-11; Primary Completion 2011-02 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
The primary purpose of this pilot study is to test the feasibility of implementing Tu Salud Si Cuenta in a worksite environment. | One year

CONTACTS AND LOCATIONS:
Overall Officials: Belinda Reininger, DrPH, Principal Investigator — University of Texas Health Science Center at Houston School of Public Health - Brownsville Regional Campus
Locations (2):
- United States (2):
  - City of Brownsville, Brownsville, Texas
  - State Department of Public Health Region 11 Harlingen Office, Harlingen, Texas

REFERENCES:
- [Background] Wang Y, Beydoun MA. The obesity epidemic in the United States--gender, age, socioeconomic, racial/ethnic, and geographic characteristics: a systematic review and meta-regression analysis. Epidemiol Rev. 2007;29:6-28. doi: 10.1093/epirev/mxm007. Epub 2007 May 17. PMID 17510091
- [Background] Wang Y, Zhang Q. Are American children and adolescents of low socioeconomic status at increased risk of obesity? Changes in the association between overweight and family income between 1971 and 2002. Am J Clin Nutr. 2006 Oct;84(4):707-16. doi: 10.1093/ajcn/84.4.707. PMID 17023695
- [Background] Wang Y, Beydoun MA, Liang L, Caballero B, Kumanyika SK. Will all Americans become overweight or obese? estimating the progression and cost of the US obesity epidemic. Obesity (Silver Spring). 2008 Oct;16(10):2323-30. doi: 10.1038/oby.2008.351. Epub 2008 Jul 24. PMID 18719634
- [Background] Craig CL, Marshall AL, Sjostrom M, Bauman AE, Booth ML, Ainsworth BE, Pratt M, Ekelund U, Yngve A, Sallis JF, Oja P. International physical activity questionnaire: 12-country reliability and validity. Med Sci Sports Exerc. 2003 Aug;35(8):1381-95. doi: 10.1249/01.MSS.0000078924.61453.FB. PMID 12900694
- [Background] Fava JL, Ruggiero L, Grimley DM. The development and structural confirmation of the Rhode Island Stress and Coping Inventory. J Behav Med. 1998 Dec;21(6):601-11. doi: 10.1023/a:1018752813896. PMID 9891257
- [Background] Finley, R. (2008). SurveyMonkey.com [Computer software]. Portland, OR: SurveyMonkey.com.
- [Background] Haskell WL, Lee IM, Pate RR, Powell KE, Blair SN, Franklin BA, Macera CA, Heath GW, Thompson PD, Bauman A. Physical activity and public health: updated recommendation for adults from the American College of Sports Medicine and the American Heart Association. Med Sci Sports Exerc. 2007 Aug;39(8):1423-34. doi: 10.1249/mss.0b013e3180616b27. PMID 17762377
- [Background] Hoelscher DM, Day RS, Kelder SH, Ward JL. Reproducibility and validity of the secondary level School-Based Nutrition Monitoring student questionnaire. J Am Diet Assoc. 2003 Feb;103(2):186-94. doi: 10.1053/jada.2003.50031. PMID 12589324
- [Background] Wolfinger, R. & O'Connell, M. (1993). Generalized linear mixed effects models: A pseudo-likelihood approach. Journal of Statistical Computation and Simulation, 48, 233-243.
- [Background] Zeger SL, Liang KY. Longitudinal data analysis for discrete and continuous outcomes. Biometrics. 1986 Mar;42(1):121-30. PMID 3719049